CLINICAL TRIAL: NCT00187681
Title: Effect of Genetic Variants in the Xenobiotic Transporter, OCT1, on Response to Metformin in Healthy Subjects
Brief Title: Organic Cation Transporter 1 (OCT1), on Response to Metformin in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 865
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2013-01-08 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2012-12

CONDITIONS: Other Conditions That May Be A Focus of Clinical Attention
Keywords: Healthy controls
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OCT1-variant Group (Experimental): Subjects with OCT1-variant alleles will be dosed with 2 doses of Metformin
  Interventions: Drug: Metformin
- OCT1-reference Group (Experimental): Subjects with OCT1-reference alleles will be dosed with 2 doses of Metformin
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 2 doses of Metformin Day 1 1000mg, Day 2 850 mg
  Other Names: Dimethylguanylguanidine; Glucophage

SUMMARY:
Specific Objectives:

* To determine if individuals who carry a decreased or non-functional variant of OCT1 exhibit differences in the pharmacokinetics of metformin in comparison to individuals who carry the common allele.
* To determine if individuals who carry the decreased or non-functional variants exhibit differences in the response to metformin in comparison to individuals who carry the common allele.

DETAILED DESCRIPTION:
In the proposed studies, we will address two questions:

•Do individuals who carry one of OCT1 variants with reduced or no function exhibit differences in the pharmacokinetics of metformin in comparison to individuals who carry the common allele?

Compared to wild type mice, Oct1-/- mice have reduced metformin distribution to the liver and intestine. We expect a similar pattern between persons who carry the variant OCT1 allele and those who carry the common allele. This effect might be reflected by a difference of Tmax or Cmax after oral administration of metformin. Other differences in metformin pharmacokinetic properties such as volume of distribution, half life and clearance may also be evident.

•Do individuals who carry the decreased or non-functional variants exhibit differences in the response to metformin in comparison to individuals who carry the common allele? Specially, we will test the hypothesis that the OCT1-expressing tissues are target organs for metformin, and that individuals with the variant transporters may have reduced metformin uptake into these sites (is this the correct meaning?) and therefore a reduced drug response to metformin.

In this study, we will evaluate metformin pharmacokinetics and glucose metabolic effects in healthy subjects rather than in patients with type 2 diabetes. Our rationale is as follows. The hepatic glucose production in diabetic patients is abnormally increased. Metformin decreases fasting blood glucose concentration by reducing hepatic glucose production and improving glucose utilization. However, the fasting blood glucose concentration is not decreased by metformin in non-diabetics who have a normal hepatic glucose production. It was suggested that the glucose-lowering effect of metformin was difficult to demonstrate in non-diabetics unless glucose concentrations were artificially raised. Although there are studies showing that metformin improves the glucose tolerance both in non-diabetics and diabetics, the results for non-diabetics have been inconsistent, depending on the variable experimental condition. Variation in OCT1 expression and activity may be one of those variables, and the time points for blood sampling after drug and glucose (meal) intakes may also be important to observe the glucose-lowering effect [16]. In this study, we employ a similar study design as that reported [16] to observe the glucose-lowering effect by metformin in healthy subjects. Before and after metformin administration, oral glucose tolerance test (OGTT) will be conducted. We expect a difference of glucose tolerance between different OCT1 genotypes, under the hypothesis that individuals with different OCT1 genotypes have different metformin concentrations in the target tissues, and hence have different glucose uptakes into (and so utilization in) the target tissues (primary muscle and liver).

In non-diabetic healthy subjects, metformin significantly attenuated the rise in immediate postprandial insulin levels. In this study, we will also determine insulin levels after glucose administration. With metformin treatment, we expect to observe significant difference in post-glucose-administration insulin levels between individuals with different OCT1 genotypes.

When mice were given metformin, the blood lactate concentration significantly increased in the wild-type mice, whereas only a slight increase was observed in Oct1-/- mice. This is consistent with our hypothesis that OCT1 is a determinant of metformin effect on glucose utilization. It will be interesting to compare plasma lactate concentrations after metformin treatment between individuals with different OCT1 genotypes.

Metformin can improve lipid metabolism in obese and diabetics patients, which is reflected by the reduced plasma levels of free fatty acid, cholesterol, and triglycerides. However, in this study with a single dose of metformin, it may not be possible to observe those effects in healthy subjects, although the corresponding concentrations will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in the Study Of Pharmacogenetics In Ethnically Diverse Populations (SOPHIE) study.
* Between the ages of 18 and 40.
* Possess a specific OCT1 genotype.

Exclusion Criteria:

* Taking any medications other than vitamins
* Individuals with anemia (hemoglobin < 12 g/dL), an elevation in liver enzymes to higher than double the respective normal value, or elevated creatinine concentrations (males ≥ 1.5 mg/dL, females ≥ 1.4 mg/dL)
* Pregnant at time of study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2003-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Giacomini, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francsico, California, United States

REFERENCES:
- [Result] Shu Y, Sheardown SA, Brown C, Owen RP, Zhang S, Castro RA, Ianculescu AG, Yue L, Lo JC, Burchard EG, Brett CM, Giacomini KM. Effect of genetic variation in the organic cation transporter 1 (OCT1) on metformin action. J Clin Invest. 2007 May;117(5):1422-31. doi: 10.1172/JCI30558. PMID 17476361
- [Result] Shu Y, Brown C, Castro RA, Shi RJ, Lin ET, Owen RP, Sheardown SA, Yue L, Burchard EG, Brett CM, Giacomini KM. Effect of genetic variation in the organic cation transporter 1, OCT1, on metformin pharmacokinetics. Clin Pharmacol Ther. 2008 Feb;83(2):273-80. doi: 10.1038/sj.clpt.6100275. Epub 2007 Jul 4. PMID 17609683

RESULTS

PARTICIPANT FLOW:
Groups:
- Organic Cation Transporter 1 (OCT1)-Variant Group: Subjects with OCT1-variant alleles to be dosed with 2 doses of Metformin (total 1850 mg).
- Organic Cation Transporter 1 (OCT1)-Reference Group: Subjects with OCT1-reference alleles to be dosed with 2 doses of Metformin (total 1850 mg).
Period: Overall Study
Arm/Group | Organic Cation Transporter 1 (OCT1)-Variant Group | Organic Cation Transporter 1 (OCT1)-Reference Group
Started | 12 | 8
Completed | 12 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- OCT1-variant Group; OCT1-reference Group: Subjects with OCT1-reference alleles to be doses with 2 doses of Metformin (total 1850 mg).
- Total: Total of all reporting groups
Arm/Group | OCT1-variant Group | OCT1-reference Group | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 8 | 20
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.0 (5.9) | 31.3 (5.4) | 30.5 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Blood Concentration-time of Metformin
Description: To test whether individuals with genetic variants of human organic cation transporter, OCT1, exhibit altered pharmacokinetics of metformin, the difference in AUC of blood concentration-time of metformin between reference and variant groups will be measured.
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, and 24 hours
Population: 20 participants were analyzed as per protocol. The sample size of 20 subjects enabled us to detect a significant difference (at the p < 0.05 level; α = 0.05, β = 0.80) in the pharmacokinetics of metformin between individuals who are homozygous for the reference OCT1 and those who carry an OCT1-R61C, OCT1-G401S or OCT1-G465R allele.
Measure: Mean (Standard Deviation); unit: hour * µg/L
Groups:
- OCT1-variant Group: Metformin blood concentration-time profiles in subjects carrying the variant OCT1 genotypes (ie. carries at least one of the four variant alleles OCT1-R61C, G401S, 420del, and/or OCT1-G465R).
- OCT1-reference Group: Metformin blood concentration-time profiles in subjects carrying the reference OCT1 allele at all the four positions in the OCT1 gene.
Arm/Group | OCT1-variant Group | OCT1-reference Group
Number analyzed (Participants) | 12 | 8
hour * µg/L | 9,200 (1,200) | 7,700 (970)

2. Primary Outcome: Glucose Lowering Response to Metformin
Description: To test whether individuals with genetic variants of human organic cation transporter, OCT1, exhibit altered glucose lowering response to metformin we will measure the difference in area under the glucose concentrations-time curve (Glucose AUC) following oral glucose tolerance test.
Time Frame: 0 to 180 minutes
Population: 20 participants were analyzed as per protocol. The sample size of 20 subjects enabled us to detect a significant difference (at the p < 0.05 level; α = 0.05, β = 0.80) in the pharmacodynamics of metformin between individuals who are homozygous for the reference OCT1 and those who carry an OCT1-R61C, OCT1-G401S or OCT1-G465R allele.
Measure: Mean (Standard Deviation); unit: min * mg/dL
Groups:
- OCT1-variant Group: Glucose lowering response to metformin (Glucose AUC) in subjects carrying variant OCT1 genotypes (ie. carries at least one of four variant alleles OCT1-R61C, G401S, 420del, and/or OCT1-G465R).
- OCT1-reference Group: Glucose lowering response to metformin (Glucose AUC) in subjects carrying the reference OCT1 genotype at all the four positions in the OCT1 gene.
Arm/Group | OCT1-variant Group | OCT1-reference Group
Number analyzed (Participants) | 12 | 8
min * mg/dL | 18,200 (1,600) | 21,300 (2,290)

ADVERSE EVENTS:
Arm/Group | OCT1-variant Group | OCT1-reference Group
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/12 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes